CLINICAL TRIAL: NCT07229664
Title: Clinical Study to Evaluate Safety and Effectiveness of Vinpocetine in Patients With Parkinsonian Disease
Brief Title: Vinpocetine in Patients With Parkinsonian Disease
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5469
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; vinpocetine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group (Levo-dopa group, n =30) who will receive levodopa/carbidopa (125/12.5 mg) three times daily for 6 months
  Interventions: Drug: Levodopa Carbidopa
- Vinpocetine group (Active Comparator): Patients will receive levodopa/carbidopa (125/12.5 mg) three times daily plus vinpocetine 10 mg three times daily for 6 months
  Interventions: Drug: Levodopa Carbidopa; Drug: Vinpocetine

INTERVENTIONS:
Drug: Levodopa Carbidopa — Carbidopa/levodopa, also known as levocarb and co-careldopa, is the combination of the two medications carbidopa and levodopa. It is primarily used to manage the symptoms of Parkinson's disease.
Drug: Vinpocetine — VIN, a phosphodiesterase-1 (PDE1) inhibitor, reduces oxidative stress and neuroinflammation and is used clinically for cerebrovascular disease and dementia. In PD, VIN increases dopamine levels, protects dopaminergic neurons, reverses motor impairments, and reduces inflammatory mediators
  Arms: Vinpocetine group

SUMMARY:
The clinical manifestations of Parkinson's disease (PD), a chronic neurodegenerative condition, include resting tremor, hypokinesia, bradykinesia, stiffness and postural instability. These motor symptoms are caused by a selective loss and degeneration of dopaminergic neurons in the substantia nigra pars compacta (SNpc) region, which leads to a dopamine (DA) insufficiency in the striatum

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 50 years Both male and female will be included Negative pregnancy test and effective contraception. Diagnosed Parkinson's disease patient taking Levodopa

Exclusion Criteria:

Secondary causes of parkinsonism Patients taking anti-inflammatory drugs Atypical parkinsonian syndromes Prior stereotaxic surgery for Parkinson's disease Pregnancy and lactation Cardiovascular disease patients Patients with coagulation disorders Suffering from active malignancy Addiction to alcohol and / or drugs Known allergy to the studied medications

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in The Unified Parkinson's Disease Rating Scale (UPDRS). | 6 months
  The unified Parkinson's disease rating scale is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease.

SECONDARY OUTCOMES:
changes in serum biomarkers | 6 months
  The secondary endpoint is estimated by changes in serum biomarkers such as α-synuclein and Toll like receptor 4

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt